CLINICAL TRIAL: NCT03309605
Title: A Phase 1, Randomized, Double-Blinded, Placebo-Controlled, Third Party Open, Multiple Dose Escalation, Single Center Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Subcutaneously Administered ELX-02 in Independent Consecutive Cohorts of Healthy Subjects
Brief Title: Phase 1 Study of ELX-02 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eloxx Pharmaceuticals, Inc. (Industry)
Collaborators: SGS Life Sciences, a division of SGS Belgium NV (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EL-002
Record Dates: First submitted 2017-10-10; First posted 2017-10-13 (Actual); Results first posted 2021-03-16 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-02

CONDITIONS: Genetic Disease; Nonsense Mutation
Keywords: Translational read through
MeSH Terms: conditions — Genetic Diseases, Inborn | interventions — ELX-02

STUDY DESIGN:
Intervention Model Description: * Cohort 1: ELX-02 0.1 mg/kg or placebo SC twice a week for 9 doses;
  * Cohort 2: ELX-02 0.3 mg/kg or placebo SC twice a week for 9 doses;
  * Cohort 3: ELX-02 1.0 mg/kg or placebo SC twice a week for 9 doses;
  * Cohort 4: ELX-02 2.5 mg/kg or placebo SC twice a week for 9 doses;
  * Cohort 5: ELX-02 up to 2.5 mg/kg (50 mg/mL per injection) or placebo SC twice a week for 9 doses;
  * Cohort 6: ELX-02 2.5 to 5.0 mg/kg or placebo SC twice a week for 9 doses. Optional Cohort
  * Cohort 7: ELX-02 up to 5.0 mg/kg or placebo SC twice a week for 9 doses. Optional Cohort
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Comparator Arm (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- ELX-02 (Experimental): ELX-02
  Interventions: Drug: ELX-02

INTERVENTIONS:
Drug: ELX-02 — ELX-02 is a synthetic, designer eukaryotic ribosomal specific glycoside (ERSG) optimized as a translational read-through drug
  Arms: ELX-02
Drug: Placebo — Placebo
  Arms: Placebo Comparator Arm

SUMMARY:
Phase 1 Multiple Ascending Dose Study in Normal Healthy Volunteers

DETAILED DESCRIPTION:
This is a study in humans of ELX-02, an advanced synthetic aminoglycoside optimized as a translational read-through drug (TRID) for the treatment of genetic conditions caused by nonsense mutations. This is a classical Phase 1b study designed as a randomized, double-blinded, placebo-controlled, multiple dose escalation to evaluate the safety, tolerability, and pharmacokinetics of ELX-02 in healthy adult volunteers.

ELIGIBILITY:
Inclusion criteria: Subjects must meet all of the following inclusion criteria to be eligible for enrollment into the study:

1. Be able and willing to provide written Informed Consent indicating that the subject has been informed of all pertinent aspects of the study.
2. Healthy female subjects and male subjects who, at the time of screening, are between the ages of 18 and 55 years, inclusive.

   Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure (BP) and pulse rate measurement, 12-lead electrocardiogram (ECG), and clinical laboratory tests.
3. Female subjects of non-childbearing potential must meet at least one of the following criteria:

   * Achieved postmenopausal status, defined as follows: cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; post-menopausal status will be confirmed by a serum follicle-stimulating hormone level;
   * Have undergone a documented hysterectomy and/or bilateral oophorectomy;
   * Have medically confirmed ovarian failure. All other female subjects (including females with tubal ligations) will be considered to be of childbearing potential and may be enrolled if they have negative pregnancy tests at screening and admission day and agree to use a highly effective method of contraception for 14 days before first study drug administration and 28 days after last study drug administration. Female subjects of childbearing potential must agree to undergo repeated pregnancy tests.
4. Male subjects must be willing to use an effective method of contraception. They must agree to use a condom consistently and correctly, during the course of the study until 28 days after last study drug administration.
5. Not using any prescription medication and dietary supplements within 30 days or 5 half lives (whichever is longer) prior to the first study drug administration, except for contraceptives - nor be taking any over-the-counter (OTC) herbal or medicinal products. As an exception, acetaminophen/paracetamol may be used at doses of ≤2 g/day.
6. Non-smoking and no use of any tobacco or nicotine products (by declaration) for a period of at least 6 months prior to screening visit.
7. Be on no medication with potential to impair renal function (e.g., non steroidal anti inflammatory [NSAID]s) or with ototoxic potential (e.g., quinine, salicylates, aminoglycosides).
8. Normal renal function (glomular filtration rate >60 mL/min) based on creatinine plasma concentration and the Modification of Diet in Renal Disease (MDRD) equation for estimated glomular filtration rate. Subjects with lower MDRD clearance can be included on the condition that they have a normal 24h creatinine clearance (determined by a 24h urine collection).
9. Negative human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) serology tests at screening.
10. No history of alcohol or DOA. Negative urine test for DOA and alcohol breath test at screening and Day -1.
11. No personal history (or current) or hereditary hearing loss, persistent tinnitus, persistent vertigo, persistent imbalance and persistent unsteadiness.
12. Body Mass Index (BMI) of 19.0 to 30.0 kg/m2 (inclusive); and a total body weight >50.0 kg (110 lbs) and <100.0 kg.

Exclusion criteria: Subjects with any of the following characteristics/conditions will not be included in the study:

1. Subjects who are investigational site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the Investigator, or subjects who are the Sponsor employees directly involved in the conduct of the study.
2. Concurrent participation or participation in another clinical trial within at least 5 tissue half-lives prior to dosing (calculated from the previous study's last dosing day). If the previous trial involved agents with delayed effects or prolonged metabolism, a 12 months interval is required.
3. Evidence or history of clinically relevant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies). This includes any acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational drug administration or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the subject inappropriate for entry into this study.
4. Presence of mitochondrial mutations making subject susceptible to aminoglycoside toxicity.
5. Subjects with any history of ear disease or surgeries, persistent dizziness or persistent tinnitus.
6. Subjects with any abnormality at screening, that indicates the presence of a vestibular pathology, conductive hearing loss or balance problem (by an ENT).

   Subjects with abnormalities in audiometry results at screening as follows: any pure-tone threshold >55 dB and/or inter-ear difference in any frequency of >20 dB.

   Dizziness Handicap Inventory (DHI)-H score>16. Tinnitus Handicap Inventory (THI)-H score >14.
7. History of regular alcohol consumption exceeding 14 drinks/week for females or 21 drinks/week for males (1 drink = 150 mL of wine or 360 mL of beer or 45 mL of hard liquor) within 6 months of screening.
8. Screening supine BP ≥ 140 mm Hg (systolic) or ≥ 90 mm Hg (diastolic), following at least 5 min of supine rest. If BP is ≥ 140 mm Hg (systolic) or ≥ 90 mm Hg (diastolic), the BP should be repeated two more times and the average of the three BP values should be used to determine the subject's eligibility.
9. Screening supine 12-lead ECG demonstrating QTc >450 msec for men and >470 msec for women, or a QRS interval >120 msec. If QTc or QRS exceed these limits, the ECG should be repeated two more times and the average of the three QTc or QRS values should be used to determine the subject's eligibility.
10. Subjects with ANY abnormalities in clinical laboratory tests at screening, considered by the study physician as clinically relevant. In particular, subjects with alanine aminotransferase (ALT), aspartate aminotransferase (AST), serum creatinine and total bilirubin ≥ 1.5 upper limit of normal will be excluded.
11. Pregnant or breastfeeding female subjects.
12. Subjects who donated blood or received blood or plasma derivatives in the three months preceding study drug administration.
13. Unwilling or unable to comply with all scheduled visits, treatment plan, laboratory tests and other study procedures and the restrictions described in this protocol.
14. Known relevant allergy to any drug and/or aminoglycosides.
15. Subjects with an inability to communicate well with the Investigators and CPU staff (e.g., language problem, poor mental development).
16. Subjects with visual impairment or inability to read and comprehend the DHI and THI scales.
17. Subjects with any acute medical situation (e.g., acute infection) within 48 hours of study start, which is considered of significance by the Investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2017-10-11 (Actual); Primary Completion 2019-06-17 (Actual); Study Completion 2019-07-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- SGS Life Sciences, Clinical Pharmacology Unit, Antwerp, Belgium

REFERENCES:
- [Result] Leubitz A, Vanhoutte F, Hu MY, Porter K, Gordon E, Tencer K, Campbell K, Banks K, Haverty T. A Randomized, Double-Blind, Placebo-Controlled, Multiple Dose Escalation Study to Evaluate the Safety and Pharmacokinetics of ELX-02 in Healthy Subjects. Clin Pharmacol Drug Dev. 2021 Aug;10(8):859-869. doi: 10.1002/cpdd.914. Epub 2021 Jan 19. PMID 33465285
- See also: Eloxx Pharmaceuticals Website — http://www.eloxxpharma.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All subjects were treated at medical clinics. The first patient was enrolled on 22 November 2017 and the last subject visit occurred on 18 July 2019.
Pre-assignment Details: Nine (9) subjects were to be randomized to receive ELX-02 or placebo at the 2:1 ratio in each cohort. However, only 8 subjects were randomized in Cohort 2. Subjects who received placebo in any of the 7 cohorts were pooled in the All Placebo group.
Groups:
- Cohort 1: 0.1 mg/kg Concentration 50 mg/mL, twice a week for 9 doses
- Cohort 2: 0.3 mg/kg Concentration 50 mg/mL, twice a week for 9 doses
- Cohort 3: 1.0 mg/kg Concentration 100 mg/mL, twice a week for 9 doses
- Cohort 4: 2.5 mg/kg Concentration 100 mg/mL, twice a week for 9 doses
- Cohort 5: 1.0 mg/kg Concentration 50 mg/mL, twice a week for 9 doses
- Cohort 6: 2.5 mg/kg Concentration 50 mg/mL, twice a week for 9 doses
- Cohort 7: 5.0 mg/kg Concentration 50 mg/mL, twice a week for 9 doses
- All Placebo: Placebo, twice a week for 9 doses
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | All Placebo
Started | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 21
Completed | 6 | 5 | 6 | 5 | 5 | 6 | 3 | 19
Not Completed | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1: 0.1 mg/kg Concentration 50 mg/mL
- Cohort 2: 0.3 mg/kg Concentration 50 mg/mL
- Cohort 3: 1.0 mg/kg Concentration 100 mg/mL
- Cohort 4: 2.5 mg/kg Concentration 100 mg/mL
- Cohort 5: 1.0 mg/kg Concentration 50 mg/mL
- Cohort 6: 2.5 mg/kg Concentration 50 mg/mL
- Cohort 7: 5.0 mg/kg Concentration 50 mg/mL
- All Placebo: 0 mg/kg
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | All Placebo | Total
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 21 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.2 (12.43) | 36.0 (8.69) | 37.7 (14.51) | 37.0 (11.26) | 37.8 (10.46) | 44.8 (11.14) | 33.5 (7.74) | 38.9 (11.16) | 38.5 (10.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 0 | 3 | 2 | 1 | 0 | 3 | 7 | 21
  Male | 1 | 5 | 3 | 4 | 5 | 6 | 3 | 14 | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 2 | 8
  White | 6 | 5 | 6 | 6 | 6 | 6 | 0 | 19 | 54
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Belgium | 6 | 5 | 6 | 6 | 6 | 6 | 0 | 18 | 53
  United States | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic Parameters - Plasma AUC0-24
Description: Day 1 Area under the curve (AUC0-24) of ELX-02 plasma concentration following the subcutaneous (SC) dose on Day 1 to 24 hours post-ose
Time Frame: Day 1: pre-dose, 15 min, 30 min, 45 min, 1h, 3h, 6h, 12h, 24h, post-dose
Population: Plasma ELX-02 exposure was generally similar following SC administration of either a 50 or 100 mg/mL final diluted injection solution strength, indicating no formulation-related differences in PK, therefore the results from Cohorts 3 and 5, and Cohorts 4 and 6 were combined.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Cohort 1: 0.1 mg/kg, twice a week for 9 doses
- Cohort 2: 0.3 mg/kg, twice a week for 9 doses
- Cohort 3 and Cohort 5: 1.0 mg/kg, twice a week for 9 doses
- Cohort 4 and Cohort 6: 2.5 mg/kg, twice a week for 9 doses
- Cohort 7: 5.0 mg/kg, twice a week for 9 doses
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 and Cohort 5 | Cohort 4 and Cohort 6 | Cohort 7
Number analyzed (Participants) | 6 | 5 | 12 | 12 | 6
ng*h/mL | 1105.126 (15.261) | 3125.484 (13.836) | 11018.22 (12.436) | 28235.823 (16.255) | 61906.528 (20.455)

2. Primary Outcome: Pharmacokinetic Parameters- Plasma AUC0-24
Description: Day 29 Area under the curve (AUC0-24) of ELX-02 plasma concentration following the subcutaneous (SC) dose on Day 29 to 24 hours post-dose
Time Frame: Day 29: pre-dose, 15 min, 30 min, 45 min, 1h, 3h, 6h, 12h, 24h, post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 and Cohort 5 | Cohort 4 and Cohort 6 | Cohort 7
Number analyzed (Participants) | 6 | 5 | 12 | 12 | 6
ng*h/mL | 1215.098 (15.431) | 3109.978 (16.601) | 10847.306 (14.098) | 29651.700 (23.223) | 54749.370 (13.770)

3. Primary Outcome: Pharmacokinetic Parameters - Plasma Cmax
Description: Day 1 Peak Plasma Concentration (Cmax) of ELX-02 following the subcutaneous (SC) dose on Day 1 to 72 hours post-dose
Time Frame: Day 1: pre-dose, 15 min, 30 min, 45 min, 1h, 3h, 6h, 12h, 24h, 36h, 48h, 72h, post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 and Cohort 5 | Cohort 4 and Cohort 6 | Cohort 7
Number analyzed (Participants) | 6 | 5 | 12 | 12 | 6
ng/mL | 284.710 (21.060) | 1003.266 (5.766) | 2880.233 (11.647) | 7721.256 (6.387) | 15912.090 (17.265)

4. Primary Outcome: Pharmacokinetic Parameters - Plasma Cmax
Description: Day 29 Peak Plasma Concentration (Cmax) of ELX-02 following the subcutaneous (SC) dose on Day 29 to 72 hours post-dose
Time Frame: Day 29: pre-dose, 15 min, 30 min, 45 min, 1h, 3h, 6h, 12h, 24h, 36h, 48h, 72h post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 and Cohort 5 | Cohort 4 and Cohort 6 | Cohort 7
Number analyzed (Participants) | 6 | 5 | 12 | 12 | 6
ng/mL | 342.779 (12.021) | 961.448 (7.460) | 2806.966 (16.403) | 7852.172 (12.342) | 15435.789 (13.872)

5. Primary Outcome: Pharmacokinetic Parameter - Plasma AUC0-inf
Description: Day 1 Area under the curve (AUC0-inf) of ELX-02 plasma concentration following the subcutaneous (SC) dose on Day 1 extrapolated to infinity
Time Frame: Day 1: pre-dose, 15 min, 30 min, 45 min, 1h, 3h, 6h, 12h, 24h, 36h, 48h, 72h post dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 and Cohort 5 | Cohort 4 and Cohort 6 | Cohort 7
Number analyzed (Participants) | 6 | 5 | 12 | 12 | 6
ng*hr/mL | 1107.272 (15.345) | 3127.964 (13.898) | 11036.305 (12.631) | 28335.680 (16.468) | 62142.763 (20.712)

6. Primary Outcome: Pharmacokinetic Parameter - Plasma AUC0-inf
Description: Day 29 Area under the curve (AUC0-inf) of ELX-02 plasma concentration following the subcutaneous (SC) dose on Day 29 extrapolated to infinity
Time Frame: Day 29: pre-dose, 15 min, 30 min, 45 min, 1h, 3h, 6h, 12h, 24h, 36h, 48h, 72h post dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 and Cohort 5 | Cohort 4 and Cohort 6 | Cohort 7
Number analyzed (Participants) | 6 | 5 | 12 | 12 | 6
ng*h/mL | 1216.448 (15.428) | 3114.486 (16.704) | 10862.927 (14.239) | 29778.143 (23.469) | 54933.538 (13.979)

7. Primary Outcome: Pharmacokinetic Parameter - Plasma Tmax
Description: Day 1 Time to maximum concentration (Tmax) of ELX-02 plasma concentrations following the subcutaneous (SC) dose on Day 1
Time Frame: Day 1: pre-dose, 15 min, 30 min, 45 min, 1h, 3h, 6h, 12h, 24h, 36h, 48h, 72h post-dose
Population: as for outcome 1
Measure: Median (Full Range); unit: hour
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 and Cohort 5 | Cohort 4 and Cohort 6 | Cohort 7
Number analyzed (Participants) | 6 | 5 | 12 | 12 | 6
hour | 1.00 [0.50 to 3.00] | 0.75 [0.50 to 1.00] | 1.00 [0.75 to 1.00] | 1.00 [0.75 to 1.00] | 0.86 [0.73 to 1.00]

8. Primary Outcome: Pharmacokinetic Parameter Plasma - Tmax
Description: Day 29 Time to maximum concentration (Tmax) of ELX-02 plasma concentrations following the subcutaneous (SC) dose on Day 29
Time Frame: Day 29: pre-dose, 15 min, 30 min, 45 min, 1h, 3h, 6h, 12h, 24h, 36h, 48h, 72h post-dose
Measure: Median (Full Range); unit: hour
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 and Cohort 5 | Cohort 4 and Cohort 6 | Cohort 7
Number analyzed (Participants) | 5 | 5 | 11 | 11 | 3
hour | 1.00 [0.50 to 1.00] | 0.75 [0.75 to 1.00] | 1.00 [0.75 to 1.00] | 0.75 [0.75 to 1.00] | 0.98 [0.73 to 0.98]

9. Primary Outcome: Pharmacokinetic Parameter - Plasma Rac(AUC24h)
Description: Accumulation ratio, calculated as AUC24h Day29/AUC24h Day 1
Time Frame: Day 1 and Day 24 hr
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 and Cohort 5 | Cohort 4 and Cohort 6 | Cohort 7
Number analyzed (Participants) | 4 | 5 | 11 | 11 | 3
Ratio | 1.093 (7.497) | 0.995 (6.622) | 0.984 (7.892) | 1.056 (14.161) | 0.911 (13.377)

10. Primary Outcome: Pharmacokinetic Parameter - Plasma RAC(Cmax)
Description: Accumulation ratio, calculated as Cmax Day29/Cmax Day 1
Time Frame: Day 1 and Day 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 and Cohort 5 | Cohort 4 and Cohort 6 | Cohort 7
Number analyzed (Participants) | 5 | 5 | 11 | 11 | 3
Ratio | 1.217 (15.278) | 0.958 (7.429) | 0.976 (12.401) | 1.018 (15.413) | 0.941 (1.262)

11. Primary Outcome: Urine Pharmacokinetics Parameter - Ae72h
Description: Day 1 Cumulative amount of unchanged drug excreted into urine (Ae72h) of ELX-02 following the subcutaneous (SC) dose on Day 1
Time Frame: Day 1: pre-dose and during 0-12h, 12-24h, 24-48h, and 48-72h post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 and Cohort 5 | Cohort 4 and Cohort 6 | Cohort 7
Number analyzed (Participants) | 6 | 5 | 12 | 12 | 6
mg | 6.702 (16.721) | 15.177 (8.524) | 58.270 (20.046) | 160.665 (11.622) | 332.467 (18.102)

12. Primary Outcome: Urine Pharmacokinetics Parameter - Ae72h
Description: Day 29 Cumulative amount of unchanged drug excreted into urine (Ae72h) of ELX-02 following the subcutaneous (SC) dose on Day 29
Time Frame: Day 29: pre-dose and during 0-12h, 12-24h, 24-48h, and 48-72h post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 and Cohort 5 | Cohort 4 and Cohort 6 | Cohort 7
Number analyzed (Participants) | 6 | 5 | 12 | 12 | 6
mg | 6.331 (28.505) | 15.021 (9.189) | 66.354 (15.505) | 162.609 (12.742) | 399.302 (14.863)

13. Primary Outcome: Urine Pharmacokinetic Parameter - Rmax
Description: Day 1 Maximum rate of urinary extraction (Rmax) of EXL-02 in each collection time interval following the subcutaneous (SC) dose on Day 1
Time Frame: Day 1: pre-dose and during 0-12h, 12-24h, 24-48h, and 48-72h post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/h
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 and Cohort 5 | Cohort 4 and Cohort 6 | Cohort 7
Number analyzed (Participants) | 6 | 5 | 12 | 12 | 6
mg/h | 1.846 (30.561) | 4.759 (6.706) | 16.132 (15.540) | 41.587 (21.200) | 69.304 (13.495)

14. Primary Outcome: Urine Pharmacokinetic Parameter - Rmax
Description: Day 29 Maximum rate of urinary extraction (Rmax) of ELX-02 in each collection time interval following the subcutaneous (SC) dose on Day 29
Time Frame: Day 29: pre-dose and during 0-12h, 12-24h, 24-48h, and 48-72h post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/h
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 and Cohort 5 | Cohort 4 and Cohort 6 | Cohort 7
Number analyzed (Participants) | 6 | 5 | 12 | 12 | 6
mg/h | 1.950 (37.938) | 5.028 (15.875) | 18.327 (23.862) | 40.607 (18.389) | 89.796 (14.725)

15. Primary Outcome: Urine Pharmacokinetics Parameter - Fe12h Day 1
Description: Percent of dose excreted (Fe) in urine on Day 1
Time Frame: 12 hours
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of drug excreted
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 and Cohort 5 | Cohort 4 and Cohort 6 | Cohort 7
Number analyzed (Participants) | 6 | 5 | 12 | 12 | 6
percentage of drug excreted | 79.572 (10.030) | 79.440 (6.178) | 76.028 (17.403) | 89.639 (9.227) | 83.362 (5.495)

16. Primary Outcome: Urine Pharmacokinetics Parameter - Fe 12h on Day 29
Description: Percent of dose excreted (Fe) in urine on Day 29
Time Frame: 12 h on Day 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of drug excreted
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 and Cohort 5 | Cohort 4 and Cohort 6 | Cohort 7
Number analyzed (Participants) | 5 | 5 | 11 | 11 | 3
percentage of drug excreted | 76.095 (14.874) | 78.398 (3.615) | 88.130 (15.218) | 88.914 (4.157) | 94.219 (7.407)

17. Primary Outcome: Urine Pharmacokinetics Parameter - CLR24h on Day 1
Description: Renal clearance on Day 1 (CLR=Ae24h/plasmaAUC24h)
Time Frame: 24 hours
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 and Cohort 5 | Cohort 4 and Cohort 6 | Cohort 7
Number analyzed (Participants) | 5 | 5 | 12 | 12 | 6
L/h | 5.871 (22.645) | 4.823 (9.834) | 5.251 (19.135) | 5.653 (22.959) | 5.331 (16.660)

18. Primary Outcome: Urine Pharmacokinetics Parameter - CLR24h
Description: Renal clearance on Day 29 (CLR=Ae24h/plasmaAUC24h)
Time Frame: 24 h
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 and Cohort 5 | Cohort 4 and Cohort 6 | Cohort 7
Number analyzed (Participants) | 5 | 5 | 11 | 11 | 3
L/h | 5.152 (29.234) | 4.784 (10.828) | 6.068 (17.200) | 5.435 (28.521) | 7.239 (7.903)

19. Secondary Outcome: Number of Patients Experiencing at Least One Treatment-Emergent Adverse Events (TEAEs)
Description: TEAEs are undesirable events not present prior to medical treatment, or an already present event that worsens either in intensity or frequency following the study treatment
Time Frame: Day 1-29
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 and Cohort 5 | Cohort 4 and Cohort 6 | Cohort 7 | All Placebo
Number analyzed (Participants) | 6 | 5 | 12 | 12 | 6 | 21
Participants
  At least 1 TEAE | 3 | 5 | 11 | 12 | 6 | 14
  Related to study drug | 1 | 5 | 10 | 12 | 6 | 9

ADVERSE EVENTS:
Time Frame: From the date of signing the consent form until Day 36
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 and Cohort 5 | Cohort 4 and Cohort 6 | Cohort 7 | All Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/5 | 0/12 | 0/12 | 0/6 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/5 | 0/12 | 0/12 | 0/6 | 0/21
Other Adverse Events (participants affected / at risk) | 3/6 | 5/5 | 11/12 | 12/12 | 6/6 | 11/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=6) | Cohort 2 (N=5) | Cohort 3 and Cohort 5 (N=12) | Cohort 4 and Cohort 6 (N=12) | Cohort 7 (N=6) | All Placebo (N=21)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 0 (0)
Hyperacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Abdominal distention (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 1 (1) | 5 (8) | 10 (23) | 12 (59) | 6 (66) | 6 (7)
Injection site discoloration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0)
Injection site induration (General disorders) | 0 (0) | 0 (0) | 3 (5) | 3 (5) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (8) | 0 (0) | 0 (0)
Injection site hematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 3 (3)
Vessel puncture site hematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site scab (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Audiogram abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 4 (4) | 2 (3) | 2 (2) | 0 (0) | 2 (2)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dysmenorrhea (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-05-29): https://cdn.clinicaltrials.gov/large-docs/05/NCT03309605/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-25): https://cdn.clinicaltrials.gov/large-docs/05/NCT03309605/SAP_001.pdf